CLINICAL TRIAL: NCT00366119
Title: Phase 4 Clinical Trial to Evaluate the Antihypertensive Efficacy and Safety of Ramiprin Tab. in Essential Hypertension
Brief Title: Safety and Efficacy of Ramipril in the Treatment of Essential Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pacific Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMN-P01
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2007-03-09 (Estimated); Status verified 2007-03

CONDITIONS: Essential Hypertension
Keywords: hypertension; ramipril; blood pressure; artery stiffness; BNP; CRP
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Ramipril

INTERVENTIONS:
Drug: Ramipril

SUMMARY:
The purpose of this study is to assess which drug is more effective of Ramiprin®(ramipril) and Tritace®(ramipril) in the Treatment of Essential Hypertension

ELIGIBILITY:
Inclusion Criteria:

* mild and moderate essential hypertension (90mmHg≤DBP≤110mmHg)

Exclusion Criteria:

* 180mmHg≤SBP
* If differences greater than 20mmHg for SBP and 10mmHg for DBP between both arms are present on 3 consecutive readings
* If differences greater than 20mmHg for SBP and 10mmHg for DBP are present on 3 consecutive readings
* impaired hepatic function
* imapaired renal function
* angioedema
* aortic valvular stenosis or obstrcutive ejection disorder
* primary hyperaldosteronism
* renal transplantation, bilateral renal artery stenosis or unilateral stenosis in a single kidney, hemodialysis
* severe respiratory disease
* congestive heart failure( New York Association functional class Ⅲ or Ⅳ)
* malignant hypertension
* labile angina pectoris or myocardial infarction in the last 3 months before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2006-06; Study Completion 2007-06

PRIMARY OUTCOMES:
Reduction of DBP(diastolic blood pressure)

SECONDARY OUTCOMES:
Reduction of SBP(systolic blood pressure)
Percentage of patients with Dcrease of BP(blood pressure)
Percentage of patients with a Normalization of BP(blood pressure)
Artery stiffness(chang of pulse wave velocity)
Left ventricular diastolic function
Change of BNP
Change of CRP

CONTACTS AND LOCATIONS:
Overall Officials: HyoSoo Kim, Ph.D in MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, 28 Yeongeon-dong, Jongno-gu, South Korea